CLINICAL TRIAL: NCT03409770
Title: Optimising the Duration of Cooling Therapy in Mild Neonatal Encephalopathy
Brief Title: Optimising the Duration of Cooling in Mild Encephalopathy
Acronym: COMET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Thayyil, Sudhin (Individual)
Collaborators: Wayne State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 241031; 37318 (Registry Identifier: CPMS (NIHR Portfolio))
Record Dates: First submitted 2018-01-10; First posted 2018-01-24 (Actual); Last update posted 2023-08-04 (Actual); Status verified 2023-08

CONDITIONS: Neonatal Encephalopathy; Hypothermia Neonatal; Magnetic Resonance Spectroscopy
MeSH Terms: interventions — Hypothermia, Induced

STUDY DESIGN:
Intervention Model Description: Therapeutic hypothermia (33 to 34 C) for 2 different durations (48, or 72 h) and usual care (normothermia)
Who Masked: Outcomes Assessor
Masking Description: MR spectroscopy analysis will be masked to the allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Usual care (No Intervention): Usual care (normothermia) arm
- Therapeutic hypothermia - 48 h (Experimental): Whole body cooling (33 to 34 C) for 48 hours
  Interventions: Other: Therapeutic hypothermia
- Therapeutic hypothermia - 72 h (Experimental): Whole body cooling (33 to 34 C) for 72 hours
  Interventions: Other: Therapeutic hypothermia

INTERVENTIONS:
Other: Therapeutic hypothermia — Whole body cooling using a servo controlled device
  Arms: Therapeutic hypothermia - 48 h; Therapeutic hypothermia - 72 h

SUMMARY:
Phase II randomised control trial of whole body cooling in mild neonatal encephalopathy.

DETAILED DESCRIPTION:
Although therapeutic hypothermia for 72 hours reduces brain injury and improves long term neurodevelopmental outcomes after moderate or severe neonatal encephalopathy, the benefits and optimal duration of cooling therapy in mild encephalopathy is not known. Adverse neurodevelopmental outcomes at 2 years occur in 16% of babies with un-treated mild neonatal encephalopathy. In the phase I of the COMET trial, we have shown that it is feasible to identify and randomise babies with mild encephalopathy, and to obtain the primary outcome (proton MR spectroscopy levels of Thalamic N-acetyl Aspartate) accurately. The phase II of the COMET trial will examine the benefits and optimal duration of cooling therapy in babies with mild encephalopathy.

Research questions

1. Does whole body cooling initiated within 6 hours of birth and continued for 72 hours increase thalamic MR spectroscopy N-acetyl aspartate levels in babies with mild encephalopathy, when compared with those who are not cooled? (Cohort 1)
2. In babies with mild encephalopathy undergoing cooling therapy as clinical care, does rewarming at 48 hours as opposed to 72 hours result in similar thalamic N-acetyl aspartate levels? (Cohort 2)

Study Population Cohort 1: A total of 60 babies with mild encephalopathy (>36 weeks; >2Kg) aged less than 6 hours will be recruited from several tertiary neonatal units in the UK, Europe, USA and Canada, over a 2 year period. The babies will be randomised to usual care (no cooling) or cooling therapy (core temperature 33 to 34 C) for 72 hours within six hours of birth. MR imaging and spectroscopy will be performed between 4 to 14 days after birth.

Cohort 2: A total of 80 babies will mild encephalopathy (>36 weeks; >2Kg) aged 24 to 48 hours and undergoing cooling therapy as a part of standard clinical care will be recruited from several UK cooling centres, over a 2 year period. The babies will be randomised to rewarming after 48 hours or 72 hours of cooling therapy. MR imaging and spectroscopy will be performed between 4 to 14 days after birth. The babies recruited to cohort 1 will not be eligible for recruitment to cohort 2.

Primary outcome (both cohorts)

• Proton MR spectroscopy Thalamic N-acetyl aspartate levels between 4 to 14 days of age.

Benefits of the trial These data will inform the national and international guidelines on management of babies with mild neonatal encephalopathy. If a shorter duration of cooling is as good or better than 3 days of cooling, this will reduce the intensive care stays, opioid use and separation from parents.

ELIGIBILITY:
INCLUSION CRITERIA

All of the following three criteria should be met:

1. Age less than six hours. AND
2. Evidence of acute perinatal asphyxia

   1. Metabolic acidosis (pH <7.0 and/or BE >-16) in cord gas or a blood gas within one of birth.

      OR
   2. If the pH or BE is borderline (pH<7.15 to 7.0) and/or BE >-10 to -16) in cord and/or blood gas within 1h of birth additional evidence of perinatal asphyxia is required, which includes either an acute obstetric event (e.g. cord prolapse, abruption, shoulder dystocia) OR Need for continued resuscitation or ventilation at 10 minutes and/or a 10 min Apgar score <6
3. Evidence of mild NE (at-least two abnormalities) on an NICHD neurological examination performed between 1 and 6h of birth.

EXCLUSION CRITERIA

The following group of babies will be excluded prior to randomisation

1. Babies without encephalopathy
2. Babies with moderate or severe encephalopathy who meet the current NICE/AAP guidelines for cooling therapy.
3. Babies with seizures (clinical and/or aEEG/EEG)
4. Babies with moderate or severe abnormalities on aEEG voltage criteria.
5. Babies with life threatening congenital malformations

Max Age: 6 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2019-10-10 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Thalamic N-acetyl aspartate level | 4 to 14 days after birth
  Feasibility of obtaining Proton MR spectroscopy thalamic N-acetyl aspartate level

SECONDARY OUTCOMES:
Brain injury on conventional MR imaging | 4 to 14 days after birth
  Cortical, white matter or deep nuclei injury
Hospital stay | Upto 30 days after birth
  Duration of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Sudhin Thayyil, PhD, Principal Investigator — Imperial College London
Locations (8):
- Wayne State University, Michigan Center, Michigan, United States
- Luigi Vanvitelli Hospital, Naples, Italy
- United Kingdom (6):
  - Birmingham Womens Hospital, Birmingham
  - Medway NHS Foundation Trust, Gillingham
  - Liverpool Womens Hospital, Liverpool
  - Homerton University Hospital, London
  - Imperial College London, London
  - The Newcastle Upon Tyne NHS Foundation Trust, Newcastle

IPD SHARING:
Plan to Share IPD: Yes
Data can be shared unconditionally will be made available when scientific manuscripts are published.
  Data that cannot be shared publicly (e.g. to protect patient confidentiality) will be by request only. The PI will review each request on case-by-case basis. Upon approval the data requester will be asked to sign a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data will be available 3 to 6 after the end of the study.
Access Criteria: Unidentified data will be shared by publication. Request for data that affects patient confidentiality will review by the study PI on a case-by-case basis.

REFERENCES:
- [Background] Prempunpong C, Chalak LF, Garfinkle J, Shah B, Kalra V, Rollins N, Boyle R, Nguyen KA, Mir I, Pappas A, Montaldo P, Thayyil S, Sanchez PJ, Shankaran S, Laptook AR, Sant'Anna G. Prospective research on infants with mild encephalopathy: the PRIME study. J Perinatol. 2018 Jan;38(1):80-85. doi: 10.1038/jp.2017.164. Epub 2017 Nov 2. PMID 29095433
- [Background] Oliveira V, Singhvi DP, Montaldo P, Lally PJ, Mendoza J, Manerkar S, Shankaran S, Thayyil S. Therapeutic hypothermia in mild neonatal encephalopathy: a national survey of practice in the UK. Arch Dis Child Fetal Neonatal Ed. 2018 Jul;103(4):F388-F390. doi: 10.1136/archdischild-2017-313320. Epub 2017 Sep 23. PMID 28942433
- [Background] Lally PJ, Montaldo P, Oliveira V, Swamy RS, Soe A, Shankaran S, Thayyil S. Residual brain injury after early discontinuation of cooling therapy in mild neonatal encephalopathy. Arch Dis Child Fetal Neonatal Ed. 2018 Jul;103(4):F383-F387. doi: 10.1136/archdischild-2017-313321. Epub 2017 Sep 21. PMID 28935718
- [Background] Lally PJ, Pauliah S, Montaldo P, Chaban B, Oliveira V, Bainbridge A, Soe A, Pattnayak S, Clarke P, Satodia P, Harigopal S, Abernethy LJ, Turner MA, Huertas-Ceballos A, Shankaran S, Thayyil S. Magnetic Resonance Biomarkers in Neonatal Encephalopathy (MARBLE): a prospective multicountry study. BMJ Open. 2015 Sep 30;5(9):e008912. doi: 10.1136/bmjopen-2015-008912. PMID 26423856
- [Background] Robertson NJ, Thayyil S, Cady EB, Raivich G. Magnetic resonance spectroscopy biomarkers in term perinatal asphyxial encephalopathy: from neuropathological correlates to future clinical applications. Curr Pediatr Rev. 2014;10(1):37-47. doi: 10.2174/157339631001140408120613. PMID 25055862
- [Background] Lally PJ, Price DL, Pauliah SS, Bainbridge A, Kurien J, Sivasamy N, Cowan FM, Balraj G, Ayer M, Satheesan K, Ceebi S, Wade A, Swamy R, Padinjattel S, Hutchon B, Vijayakumar M, Nair M, Padinharath K, Zhang H, Cady EB, Shankaran S, Thayyil S. Neonatal encephalopathic cerebral injury in South India assessed by perinatal magnetic resonance biomarkers and early childhood neurodevelopmental outcome. PLoS One. 2014 Feb 5;9(2):e87874. doi: 10.1371/journal.pone.0087874. eCollection 2014. PMID 24505327
- [Background] Thayyil S, Chandrasekaran M, Taylor A, Bainbridge A, Cady EB, Chong WK, Murad S, Omar RZ, Robertson NJ. Cerebral magnetic resonance biomarkers in neonatal encephalopathy: a meta-analysis. Pediatrics. 2010 Feb;125(2):e382-95. doi: 10.1542/peds.2009-1046. Epub 2010 Jan 18. PMID 20083516
- [Derived] Montaldo P, Cirillo M, Burgod C, Caredda E, Ascione S, Carpentieri M, Puzone S, D'Amico A, Garegrat R, Lanza M, Moreno Morales M, Atreja G, Shivamurthappa V, Kariholu U, Aladangady N, Fleming P, Mathews A, Palanisami B, Windrow J, Harvey K, Soe A, Pattnayak S, Sashikumar P, Harigopal S, Pressler R, Wilson M, De Vita E, Shankaran S, Thayyil S; COMET Trial Group. Whole-Body Hypothermia vs Targeted Normothermia for Neonates With Mild Encephalopathy: A Multicenter Pilot Randomized Clinical Trial. JAMA Netw Open. 2024 May 1;7(5):e249119. doi: 10.1001/jamanetworkopen.2024.9119. PMID 38709535